CLINICAL TRIAL: NCT03336723
Title: Inflammation and Microbiology Pattern on Two-piece Zirconia Dental Implant Compared to Titanium Dental Implants. Randomized Clinical Control Trial
Brief Title: Two-Piece Zirconia Dental Implant vs Two-Piece Titanium Dental Implant- Randomized Clinical Control Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Implantology Institute (Other)
Responsible Party: Principal Investigator, Andre Chen, DMD, Implantology Institute
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: II10
Record Dates: First submitted 2017-11-05; First posted 2017-11-08 (Actual); Last update posted 2017-11-08 (Actual); Status verified 2017-11

CONDITIONS: Osseointegration Failure of Dental Implant Due to Infection; Osseointegration Failure of Dental Implant Prior to Intentional Prosthetic Loading
MeSH Terms: interventions — Dental Implants

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Two piece zirconia dental implants place subcrestally with a healing abutment at baseline (T0) and rehabilitated with a zirconia dental crown T3 3 Measures on the IL1b and IL6 at T0 baseline , T2 2 month and T3 at crown placement.Microbiological samples at T2 and T3.
  Interventions: Device: Dental Implant
- Control Group (Active Comparator): Two piece titanium dental implants place subcrestally with a healing abutment at baseline (T0) and rehabilitated with a zirconia dental crown T3 3 Measures on the IL1b and IL6 at T0 baseline , T2 2 month and T3 at crown placement.Microbiological samples at T2 and T3.
  Interventions: Device: Dental Implant

INTERVENTIONS:
Device: Dental Implant — Place a two piece zirconia dental implant on a healed ridge. At baseline, two month and crown placement take fluid samples with adsorbent paper in the per- implant crevicular fluid. At t2 and t3 repeat sample taken

SUMMARY:
2 Arms (60 subjects - 30 each arm). Experimental group with two-pice zirconia dental implant and Control group with two-piece titanium dental implant Evaluate Changes in inflammatory and microbiology levels from T0 (baseline) T2 (8 weeks) and T3 (after crown placement) Also evaluate secondary outcomes: marginal bone loss (MBL), gingival height (GH) levels, osseointegration, gender, age, time of surgery, anatomical position and implant stability. p values<0.05 were considered statistically significant

ELIGIBILITY:
Inclusion Criteria:

Single implants in any area (maxillary and mandibular), extracted teeth for at least 3 months before implant placement, with bone volumes sufficient (at least 2 mm mesial, distal, buccal and palatal) to accommodate dental implant without the need for regeneration. Controlled oral hygiene, absence of any lesions in the oral cavity, at least 2 mm keratinized tissue. In addition, patients must agree to participate in a postoperative control program and signed the informed consent.

Exclusion Criteria:

1 - allergic to local anaesthetics, or any of the other components. 2 - Patients with hepatic or renal dysfunction 3 - Patients with epilepsy, shock, cardiac conduction disorders or myasthenia gravis 4 - Patients with myocardial injury 5 - Hyperthyroidism 6 - Severe Hypertension 7 - Insufficient bone volume 8 - Smoking more than five cigarettes / day 9 - Excessive alcohol consumption 10 - localized anti-tumour radiation therapy of the oral cavity 11 - Chemotherapy 12 - Liver Diseases 13 - immunosuppressed patients 14 - Patients taking corticosteroids 15 - Pregnancy 16 - inflammatory and autoimmune diseases of the oral cavity

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-01-01 (Estimated); Primary Completion 2018-08-01 (Estimated); Study Completion 2019-01-01 (Estimated)

PRIMARY OUTCOMES:
Osseointegration | from T0 to T2 - 2 month
  measure if the healing process of bone was successful
Marginal bone loss | 4 month after T0
  measure bone level from T0 baseline to T3
IL1b concentration | 4 month
  Measure IL fluid at T0 and T2 for IL1b characterization
IL6 concentration | 4 month
  Measure IL fluid at T0 and T2 for IL1b characterization
Microbiologic samples | 4 month
  Measure crevicular fluid at T0 and T2 for bacteria characterization

IPD SHARING:
Plan to Share IPD: No